CLINICAL TRIAL: NCT02438007
Title: ARMOR3-SV: A Phase 3, Randomized, Open Label, Multi-Center, Controlled Study of Galeterone Compared to Enzalutamide in Men Expressing Androgen Receptor Splice Variant-7 mRNA (AR-V7) Metastatic (M1) Castrate Resistant Prostate Cancer (CRPC)
Brief Title: A Study of Galeterone Compared to Enzalutamide In Men Expressing Androgen Receptor Splice Variant-7 mRNA (AR-V7) Metastatic CRPC
Acronym: ARMOR3-SV
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: LTN PHARMACEUTICALS, INC. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ARMOR3-SV
Record Dates: First submitted 2015-03-19; First posted 2015-05-08 (Estimated); Last update posted 2023-03-15 (Actual); Status verified 2017-09

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — 3-hydroxy-17-(1H-benzimidazole-1-yl)androsta-5,16-diene; enzalutamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Galeterone (Experimental)
  Interventions: Drug: Galeterone
- Enzalutamide (Active Comparator)
  Interventions: Drug: Enzalutamide

INTERVENTIONS:
Drug: Galeterone — 2550 mg galeterone tablets once daily PO
  Other Names: TOK-001
  Arms: Galeterone
Drug: Enzalutamide — 160 mg enzalutamide capsules once daily PO
  Other Names: Xtandi®
  Arms: Enzalutamide

SUMMARY:
The purpose of this study is to compare galeterone to enzalutamide in men expressing androgen receptor spice variant-7 mRNA (AR-V7) in metastatic (M1) castrate resistant prostate cancer (CRPC).

ELIGIBILITY:
Inclusion Criteria:

* Progressive metastatic (M1) disease on androgen deprivation therapy
* Detectable AR-V7 from circulating tumors (CTCs)
* ECOG performance status 0 or 1

Exclusion Criteria:

* Prior treatment with second generation anti-androgens (e.g. abiraterone, enzalutamide)
* Prior treatment with chemotherapy for CRPC

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 953 (Actual)
Dates: Start 2015-06; Primary Completion 2016-07 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Radiographic Progression-free survival | ≥ 8 months

SECONDARY OUTCOMES:
Overall Survival | ≥ 8 months
Time to Initiation of Cytotoxic Chemotherapy | ≥ 8 months

OTHER OUTCOMES:
Skeletal-related Events | ≥ 8 months
Safety measured by clinical safety laboratories and adverse events | ≥ 8 months
Prostate Specific Antigen (PSA) Response ≥ 50% | ≥ 8 months
Time to PSA progression | ≥ 8 months
Time to ECOG deterioration | ≥ 8 months
Best Overall Response by RECIST 1.1 | ≥ 8 months

CONTACTS AND LOCATIONS:
Locations (117):
- United States (51):
  - Pinnacle Oncology Hematology, Scottsdale, Arizona
  - University Of Arizona Cancer Center, Tucson, Arizona
  - City of Hope, Duarte, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Prostate Oncology Specialists, Inc., Marina del Rey, California
  - UC Davis Cancer Center, Sacramento, California
  - San Bernardino Urological Associates, San Bernardino, California
  - Urology Speciality Group, Torrance, California
  - University of Colorado Cancer Center Anschultz Cancer Pavilion, Aurora, Colorado
  - The Urology Center of Colorado, Denver, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Sibley Memorial Hospital, Washington D.C., District of Columbia
  - Boca Raton Community Hospital, Inc., Boca Raton, Florida
  - University of Florida Health Cancer Center, Orlando, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - First Urology, Jeffersonville, Indiana
  - Tulane Medical Center, New Orleans, Louisiana
  - Regional Urology, LLC, Shreveport, Louisiana
  - University of Maryland Greenenbaum Cancer Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Walter Reed National Military Medical Center, Bethesda, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan Health System, Ann Arbor, Michigan
  - Karmanos Cancer Center, Detroit, Michigan
  - Urology Cancer Center and GU Research Network, Omaha, Nebraska
  - Coastal Urology Associates, Brick, New Jersey
  - Brooklyn Urology Research Group, Brooklyn, New York
  - Advanced Urology Centers of New York, Plainview, New York
  - Premier Medical Group of the Hudson Valley, Poughkeepsie, New York
  - Associated Medical Professionals of NY, Syracuse, New York
  - University of North Carolina Lineberger Cancer Center, Chapel Hill, North Carolina
  - Carolina Urology Partners, PLLC, Charlotte, North Carolina
  - Carolina Urology Partners, Concord, North Carolina
  - The Urology Group, Cincinnati, Ohio
  - Clinical Research Solutions, Middleburg Heights, Ohio
  - Oregon Urology Institute, Springfield, Oregon
  - Lancaster Urology, Lancaster, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - UPMC Cancer Centers, Pittsburgh, Pennsylvania
  - Carolina Urologic Research Center, Myrtle Beach, South Carolina
  - Urology Associates Clinical Research, Nashville, Tennessee
  - Urology Clinics of North Texas, Dallas, Texas
  - Texas Oncology/Baylor University Medical Center, Dallas, Texas
  - Urology San Antonio, San Antonio, Texas
  - Virginia Urology, Richmond, Virginia
  - Urology of Virginia, Virginia Beach, Virginia
  - The University of Wisconsin Paul P. Carbone Comprehensive Cancer Center, Madison, Wisconsin
- Australia (13):
  - St. George Private Hospital, Oncology Day Care Centre, Kogarah, New South Wales
  - Ashford Cancer Centre/Adelaide Cancer Centre Research, Kurralta Park, New South Wales
  - North Coast Cancer Institute, Port Macquarie, New South Wales
  - Prince of Wales Hospital, Randwick, New South Wales
  - Macquarie University, Sydney, New South Wales
  - Peninsula Specialist Centre, Kippa-Ring, Queensland
  - ICON Cancer Care, Southport, Queensland
  - Princess Alexandra Hospital, Woolloongabba, Queensland
  - Ashford Cancer Centre/Adelaide Cancer Centre Research, Kurralta Park, South Australia
  - Box Hill Hospital, Box Hill, Victoria
  - Monash Medical Centre, East Bentleigh, Victoria
  - Peter MacCallum Cancer Centre, East Melbourne, Victoria
  - Cabrini Hospital, Malvern, Victoria
- Belgium (4):
  - Jules Bordet Institute Clinique d'Oncologie Medicale, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Jessa Ziekenhuis, Hasselt
  - CHU Sart Tilman, Liège
- Canada (7):
  - British Columbia Cancer, Kelowna, British Columbia
  - British Columbia Cancer, Vancouver, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario
  - Princess Margaret Hospital, Toronto, Ontario
  - Centre Hospitalier De I'Universite de Montreal, Montreal, Quebec
  - Centre Hospitalier Universitaire de Quebec, Québec, Quebec
- France (13):
  - Centre Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Service de Médecine Interne Onco-Hématologie, La Roche-sur-Yon
  - Clinique Victor Hugo Centre Jean Bernard, Le Mans
  - Centre Léon Bérard, Lyon
  - Hôpital Edouard Herriot, Lyon
  - Centre Antoine Lacassagne, Nice
  - Centre René Gauducheau, Saint-Herblain
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Institut de Cancerlogie de la Loire, Saint-Priest-en-Jarez
  - Institut Gustave-Roussy, Villejuif
- Italy (7):
  - Centro Oncologico c/o Presidio Ospedaliero San Donato - Arezzo, Arezzo
  - Unità Operativa di Oncologia Ospedale Civile degli Infe, Faenza (RA)
  - Romagnolo per lo Studio e la Cura dei Tumori IRST-IRCCS - Oncologia medica, Meldola (FC)
  - AOU "S. Luigi", SCDU Oncologia Medica, Orbassano (Torino)
  - Az. Ospedaliera San Camillo-Forlanini, Roma
  - University of Turin, Torino
  - Santa Chiara Hospital, Trento
- Spain (12):
  - Hospital Clínic i Provincial de Barcelona-Oncology, Barcelona
  - Instituto Catalan de Oncologia (Hospital Durans i Reynals), Barcelona
  - Hospital General Universitario de Elche, Elche
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Spanish National Cancer Research Centre, Madrid
  - Fundación Althaia Manresa, Manresa
  - Unidad Cnio Ibima de Investigacion en Prostata, Málaga
  - Hospital Son Espases - Oncología, Palma de Mallorca
  - Hospital Clinico Universitario de Navarra, Pamplona
  - Consorci Hospitalari de Parc Taulí, Sabadell
  - Hospital Universitario Virgen del Rocio, Seville
  - IVO-Oncología Médica, Valencia
- United Kingdom (10):
  - CR-UK Institute for Cancer Studies, Birmingham, England
  - Sussex Cancer Centre, Brighton, England
  - University College of London Hospitals, London, England
  - Guy's and St. Thomas' NHS Foundation Trust, London, England
  - Southampton General Hospital, Southampton, England
  - University of Surrey Post Graduate Medical Hospital, Surrey, England
  - Royal Marsden Hospital, Surrey, England
  - The Royal Cornwall Hospital, Truro, England
  - The Beatson West of Scotland Cancer Centre, Glasgow, Scotland
  - Velindre Hospital, Cardiff, Wales

REFERENCES:
- [Derived] Aragon-Ching JB. The promising role of poly(ADP-ribose) polymerase inhibitors in prostate cancer. Asian J Androl. 2016 Jul-Aug;18(4):592-3. doi: 10.4103/1008-682X.172821. PMID 26908063